CLINICAL TRIAL: NCT07386795
Title: The Efficacy and Safety of Microbiota Transplantation Combined With Prebiotics for Treatment of Functional Constipation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Institute of Process Engineering, Chinese Academy of Sciences (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I-25PJ3047
Record Dates: First submitted 2026-01-27; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Constipation - Functional; Chronic Constipation; Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fecal Microbiota Transplantation (FMT) combined with Prebiotics (Experimental): Participants will receive a "co-localization" intervention combining Fecal Microbiota Transplantation (FMT) and prebiotics. The FMT graft is derived from screened healthy donors and processed to ensure a total viable bacterial count of ≥ 2.5×10¹² CFU. Before administration, the microbiota is physically mixed and resuspended with the prebiotic preparation according to standard procedures to enhance colonization and metabolic function.
  Interventions: Procedure: FMT

INTERVENTIONS:
Procedure: FMT — In this group, antibiotics are administered for 3 days prior to the procedure. A colonoscopy is performed, and a catheter is placed in the ileocecal region. Bacterial infusion is performed for 3 days with 100 mL graft per day. The graft is prepared using a "co-localization" strategy: before infusion, the microbiota is physically mixed and resuspended with the prebiotic preparation according to standard procedures. Blood and stool samples are collected before and after fecal microbiota transplantation (FMT), and researchers conduct follow-up evaluations of the patients' abdominal symptoms and signs.

SUMMARY:
Chronic constipation is a common gastrointestinal disorder with a global prevalence of approximately 15%, severely impacting daily life and quality of life. It also increases the mortality rate from hypertension, cardiovascular diseases, and ischemic stroke, and is closely related to the incidence of colorectal cancer, making it a major chronic disease that seriously threatens people's health and quality of life. With the increasing aging population and lifestyle factors such as sedentary behavior and low-fiber diets, the incidence of functional constipation is gradually rising. Traditional treatment of chronic constipation mainly relies on various types of laxatives, which have significant side effects with long-term use and relatively high treatment costs, while surgical treatment has limited patient acceptance. Gut microbiota is closely related to intestinal motility, and patients with chronic constipation often have gut microbiota dysbiosis, with significant differences in gut microbiota diversity and colonic mucosal microbiota structure compared to healthy individuals. In recent years, more and more studies have found that intestinal microbiota-based therapies such as probiotics, prebiotics, synbiotics, postbiotics, and fecal microbiota transplantation (FMT) can effectively prevent and treat chronic constipation. FMT, as a method to reshape the gut microbiota, has been widely used in many centers at home and abroad, for diseases including inflammatory bowel disease, irritable bowel syndrome, autism, and obesity. The overall adverse reaction rate in clinical applications is approximately 3%, mainly consisting of abdominal discomfort (bloating, abdominal pain), diarrhea, and secondary intestinal infections or even bacteremia (rare). Our center has established a fecal microbiota transplantation center at Beijing Sixth Hospital within our medical alliance. We have currently performed nearly 100 cases of FMT for the treatment of IBD, autism, functional bowel diseases, and other metabolic diseases, with a clinical efficacy rate of 64-85% for functional constipation and constipation-predominant irritable bowel syndrome. This project aims to validate an intervention strategy combining fecal microbiota transplantation (FMT) with prebiotics primarily composed of high dietary fiber, based on the theoretical framework developed by the team led by Diwei Zheng at the Institute of Process Engineering, Chinese Academy of Sciences.The team found that the core microbiota playing a major role in the FMT process determines the therapeutic efficacy of FMT on diseases.These core microbial communities can produce acetic acid and butyric acid, which are important metabolites that not only reduce inflammatory levels and improve intestinal barrier function, but also provide energy for intestinal epithelial cells. Additionally, they effectively limit the growth of opportunistic pathogens by acidifying the intestinal environment, exerting antibacterial effects, and utilizing niche effects.Therefore, when the core microbiota occupies a dominant ecological niche in the gut, the gut microbiota can support health from multiple aspects including nutrition, immunity, metabolism, and psychology. Prebiotics designed based on the characteristics of the core microbiota can significantly enhance the activity and colonization of the core microbiota.This study aims to reconstruct a healthy intestinal ecosystem through FMT and prebiotics. Simultaneously, it proposes a "co-localization" strategy, which involves physically mixing prebiotics with core microbiota during transplantation to coexist synergistically. This approach enhances the metabolic function of core microbiota more efficiently locally, promotes the production of key metabolites such as acetic acid and butyric acid, and improves the intestinal microenvironment.Compared with the traditional stepwise model of 'microbiota transplantation + prebiotic intervention', this approach can significantly reduce the dosage of prebiotics, thereby further enhancing the safety and tolerability of the intervention.This clinical study is designed as an open-label, single-arm trial, aiming to enroll 19 patients with refractory functional constipation to receive "core microbiota transplantation based on co-localization".The study will focus on evaluating the therapeutic efficacy of the treatment in improving constipation symptoms, systematically assessing its safety, and comprehensively evaluating the level of gut microbiota remodeling through microbiome and metabolome approaches.The implementation of this project will provide clinical evidence for exploring the application of core microbiota therapy in functional bowel disorders such as constipation, and lay the foundation for optimizing and promoting microecological intervention strategies.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with functional constipation (FC) according to Rome IV criteria.
* Symptoms persisting for at least 6 months, with criteria met for the last 3 months.
* Ineffective response to traditional treatments (dietary intervention, at least 2 types of laxatives, or probiotics).
* Willing to discontinue other constipation medications, herbal medicines, or supplements during the study.

Exclusion Criteria:

* History or clinical evidence of mechanical bowel obstruction (e.g., tumor or hernia).
* Diagnosis of megarectum, megacolon, or pseudo-obstruction.
* Organic intestinal abnormalities (obstruction, stenosis, cancer) or inflammatory bowel disease (IBD).
* Progressive colorectal polyps requiring treatment.
* History of gastrointestinal or abdominal surgery within the past 3 months.
* Severe cardiovascular or cerebrovascular diseases.
* Clinically significant liver function abnormalities (ALT/AST > 2x ULN, TBIL ≥ 1.5x ULN).
* Pregnancy, lactation, or planning to conceive during the study.
* Inability to undergo colonoscopy or catheter placement.
* Participation in other clinical trials within the past 3 months.
* Other health conditions deemed unsuitable by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in complete spontaneous bowel movements (CSBM) | 4 weeks
  Effect of FMT combined with prebiotics preparation on the change in complete spontaneous bowel movements (CSBM) of refractory functional constipation

SECONDARY OUTCOMES:
Frequency of SBM and CSBM | Baseline through Week 8
  Number of Spontaneous Bowel Movements (SBM) and Complete Spontaneous Bowel Movements (CSBM) per week.
Bristol Stool Form Scale (BSFS) Score | Baseline through Week 8
  Assessment of stool consistency using the BSFS (scale 1-7).
Patient Assessment of Constipation Symptoms Score | Baseline, Week 4, and Week 8
  Self-evaluation of constipation symptom severity.
Colonic Transit Time | Baseline and Week 4
  Assessed by colonic transit test to evaluate intestinal motility.
Fecal Water Content and Microbiota Composition | Baseline, Week 4, and Week 8
  Measurement of fecal water percentage and analysis of gut microbiota structure.
Incidence of Adverse Events | From enrollment through Week 8
  Number of participants with adverse events (e.g., bloating, infection).

CONTACTS AND LOCATIONS:
Overall Officials: Jingnan Li, MD, Ph.D, Study Chair — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No